CLINICAL TRIAL: NCT06057220
Title: Investigation of Immune Pathways and Microbiome Disruption as Drivers of Mutagenesis in Oesophagogastric Cancer
Brief Title: IMaC - Immune Pathways in Oesophagogastric Cancer
Acronym: IMaC
Status: Not yet recruiting | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5791
Record Dates: First submitted 2023-06-08; First posted 2023-09-28 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Oesophagogastric Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Saliva
  * Buccal mucosa swabs
  * OG mucus
  * OG mucosal biopsies
  * Gastric fluid
  * Surgically resected specimens of primary OG tumours
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Adult patients referred for oesophago-gastro-duodenoscopy (OGD) to investigate any of the following symptoms: difficulty swallowing, vomiting, reflux, anaemia, gastrointestinal (GI) bleeding, upper abdominal pain and weight loss.
  Interventions: Other: No intervention sample collection only
- Group 2: Adult patients with known BO who are undergoing OGD for surveillance
  Interventions: Other: No intervention sample collection only
- Group 3: Adult patients who have been diagnosed with OGc (Ac or SCc) and are having further investigations as part of the disease staging process such as a staging laparoscopy or further OGD
  Interventions: Other: No intervention sample collection only
- Group 4: Adult patients with OGc (Ac or SCc) who are having surgical resection of the cancer
  Interventions: Other: No intervention sample collection only

INTERVENTIONS:
Other: No intervention sample collection only — No intervention

SUMMARY:
The number of cases of oesophagogastric cancer is increasing every year. Currently, only 39% of patients with oesophageal cancer can have potentially curative treatment by the time they are diagnosed. This is because it typically presents late, and it is only when patients start to develop symptoms of advanced disease such as difficulty swallowing and weight loss, that they seek medical attention.

There are approximately 9300 new cases of oesophageal cancer in the UK each year and at 17%, it has the 5th poorest 5-year survival of all cancers in the UK.

It is diagnosed by carrying out a camera test called a gastroscopy which allows a biopsy of the cancer to be taken. This is an invasive procedure, and unlike for other types of cancer, such as bowel cancer, there is no test to risk-stratify patients at an earlier stage. Risk-stratification enables patients more likely to develop oesophagogastric cancer to be identified, which allows them to have more focused follow-up. This can potentially enable cancer to be diagnosed earlier, before the disease becomes more advanced, allowing patients to have potentially curative treatment.

Scientific research has identified that the healthy bacteria in the oesophagus and stomach changes as oesophagogastric cancer develops. The investigators want to see if similar changes can be identified in the healthy bacteria in the mouth which could be indicative of cancer developing in the oesophagus or stomach. The investigators then hope to use this information to develop a non-invasive risk-stratification tool that can be used to diagnose oesophagogastric cancer earlier and thereby enable more patients to be cured.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the interplay between immune pathways, the mucosal barrier and microbiome in oesophagogastric cancer, with the intention of identifying biologically-plausible biomarkers implicated in oesophagogastric carcinogenesis. The long-term translational objective of this work is to develop a non-invasive risk-stratification test with the aim of identifying patients at risk of developing, or with possible early oesophagogastric cancer, who can then undergo diagnostic testing with the intention of identifying early, potentially curable disease.

In order to do this, a deep understanding of the microbiome, the immune pathways, and ensuing changes at the level of the oesophagogastric mucosa is required. This work aligns with one of the cornerstones of improving survival in OGc; early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients >16 years old
2. Referred for oesophago-gastro-duodenoscopy (OGD) to investigate any of the following;

   1. Symptoms including difficulty swallowing, vomiting, reflux symptoms including heartburn, anaemia, GI bleeding, upper abdominal pain and weight loss.
   2. Oesophagitis, gastritis or GORD.
   3. Barrett's oesophagus (BO) requiring surveillance or endoscopic therapy.
3. Histologically confirmed OGc undergoing further investigation as part of staging such as laparoscopy and OGD or undergoing surgical resection (oesophagectomy/gastrectomy) as part of their treatment.

Exclusion Criteria:

1. Cancers other than adenocarcinoma or squamous cell carcinoma, including but not limited to gastro-intestinal stromal tumours (GIST), mucosa associated lymphoid tissue lymphoma (MALT lymphoma) and carcinoid tumours.
2. Patients with recurrent OGc.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Group 1 - Adult patients referred for oesophago-gastro-duodenoscopy (OGD) to investigate any of the following symptoms: difficulty swallowing, vomiting, reflux, anaemia, gastrointestinal (GI) bleeding, upper abdominal pain and weight loss.
  2. Group 2 - Adult patients with known BO who are undergoing OGD for surveillance.
  3. Group 3 - Adult patients who have been diagnosed with OGc (Ac or SCc) and are having further investigations as part of the disease staging process such as a staging laparoscopy or further OGD.
  4. Group 4 - Adult patients with OGc (Ac or SCc) who are having surgical resection of the cancer.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Derive biomarker(s) from the oropharyngeal microbiome and mucin profiles in each patient cohort | Through study completion (an average of 3 years)
  Identification of a novel biomarker detectable in salivary samples or buccal swabs from the oropharynx, that can be used as a marker of downstream neoplastic changes leading to oesophagogastric carcinoma.

SECONDARY OUTCOMES:
Characterise and compare the microbiome and mucin profiles of the oropharynx | Through study completion (an average of 3 years)
  Profile the oropharyngeal microbiome and mucin perturbations occurring across the spectrum of pre-malignant oesophgagogastic disease (Barrett's Oesophagus) and oesophagogastric cancers, including controls with no endoscopic evidence of upper Gastrointestinal (GI) pathology i.e. a normal upper GI tract, negative Helicobacter pylori tests and patients with GORD
Determine concomitant alterations in mucosal immune pathways and mucus biology | Through study completion (an average of 3 years)
  Comprehensive understanding of altered immune pathways driving oesophageal cancer and their relation to microbiota and mucus perturbations to provide targets for mechanistic investigation within experimental models
Establish causation between microbiome/immune/mucin perturbation and carcinogenesis. | Through study completion (an average of 3 years)
  Gain understanding of key pathways driving oesophageal carcinogenesis, insights that are essential for developing robust biologically-plausible early biomarkers with high clinical predictive value, through the use of in vitro models

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Royal Surrey County Hospital, Guildford
  - St Georges University Hospital, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No